CLINICAL TRIAL: NCT04721132
Title: An Open-Label, Phase II, Pre-Operative Study of Atezolizumab Plus Bevacizumab for Resectable Hepatocellular Carcinoma
Brief Title: Atezolizumab and Bevacizumab Before Surgery for the Treatment of Resectable Liver Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0791; NCI-2020-13744 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0791 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-01-07; First posted 2021-01-22 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Resectable Hepatocellular Carcinoma; Stage I Hepatocellular Carcinoma AJCC v8; Stage IA Hepatocellular Carcinoma AJCC v8; Stage IB Hepatocellular Carcinoma AJCC v8; Stage II Hepatocellular Carcinoma AJCC v8
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — atezolizumab; Bevacizumab; Immunoglobulin G; Disulfides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (atezolizumab, bevacizumab) (Experimental): Patients receive atezolizumab IV over 30-60 minutes and bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 21 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity. Patients then undergo surgery during week 12.
  Interventions: Biological: Atezolizumab; Biological: Bevacizumab; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Biological: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG7446; RO5541267; Tecentriq
Biological: Bevacizumab — Given IV
  Other Names: Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab awwb; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar GB-222; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar Mvasi; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; Bevacizumab Biosimilar Zirabev; Bevacizumab-awwb; Bevacizumab-bvzr; BP102; BP102 Biosimilar; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Mvasi; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501; Zirabev
Procedure: Therapeutic Conventional Surgery — Undergo surgery

SUMMARY:
This phase II trial studies the effect of atezolizumab and bevacizumab before surgery in treating patients with liver cancer that can be removed by surgery (resectable). Immunotherapy with monoclonal antibodies, such as atezolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Bevacizumab is a monoclonal antibody that may interfere with the ability of tumor cells to grow and spread. Giving the combination of atezolizumab and bevacizumab may help to prevent liver cancer from returning after surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

1. To evaluate safety and tolerability of atezolizumab plus bevacizumab combination therapy in the pre-operative setting.
2. To assess the rate of pathologic complete response.

SECONDARY OBJECTIVE:

To evaluate the correlation between rate of pathologic complete response, overall response rate at time of surgery (per Response Evaluation Criteria in Solid Tumors [RECIST] 1.1 and modified RECIST 1.0), duration of response as defined by time to recurrence/recurrence-free survival, in addition to overall survival.

EXPLORATORY OBJECTIVES:

1. Evaluate the predictive value of dynamic changes in fibrosis stage. Fibrosis stage will be assessed by histology by on serial tissue samples collected at baseline and at time of surgery (at 12 weeks after treatment begins).
2. To measure baseline and longitudinal changes of immune infiltration including CD8/Treg ratio and CD68+ density.
3. To explore the association between PD-L1 (and PD-L2) expression by immunohistochemistry, RNA seq genomic profiling, and antitumor efficacy
4. To evaluate baseline and longitudinal changes of tumor-necrosis factor (TNF)-α, pSTAT3, and c- MET; immune cell density such as frequency of PD-1+4-1BB+ CD8 T cells, pro-inflammatory cytokines, and hepatic fibrosis markers (APRI, FIB-4, hyaluronic acid, FibroTest [FibroSure]), non- alcoholic-fatty-liver-disease (NAFLD) fibrosis score (NFS), and enhanced liver fibrosis test (ELF)] as biomarkers of response to therapy.
5. To assess the impact of therapy on the diversity of the tumor-specific T-cell repertoire
6. To explore the correlation between immunological and molecular changes in tumor tissues and peripheral blood with TTP, time to recurrence, OS, and rate of AEs. In particular, we will evaluate the potential of pre-treatment CD8 T-cell density, PD-L1 expression, and CD68 to CD8 ratio or circulating CD68+DR-/low density to predict responsiveness to checkpoint blockade.

OUTLINE:

Patients receive atezolizumab intravenously (IV) over 30-60 minutes and bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 21 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity. Patients then undergo surgery during week 12.

After completion of study treatment, patients are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Must provide written informed consent prior to initiating any trial related procedures.
2. Patient must be ≥ 18 years of age
3. Patient has histologically confirmed (if tumor tissue is unavailable, documentation of diagnosis from original biopsy is acceptable) or clinically diagnosed (American Association for the Study of Liver Disease criteria in cirrhotic subjects) hepatocellular carcinoma (HCC).
4. Patient has resectable disease with no evidence of extrahepatic spread. The determination of resectability status will ultimately lie in the clinical judgment of the surgical oncologist and medical oncologist involved in the care of the patient.
5. Must have a Child-Turcotte-Pugh score of A
6. Patients must have at least one measurable site of disease per RECIST version 1.1(Appendix 4) or Immune- Modified RECIST. This is defined as a lesion that can be accurately measured in at least one dimension and measures a minimum of ≥ 10 mm (longest diameter to be recorded) with US, MRI or Spiral CT.
7. Patient has record of treated (as necessary per local SoC guidelines) or absent esophageal varices by esophagogastroduodenoscopy within 6 months of initiating treatment.
8. Patient must be willing to undergopretreatment research biopsy to provide a tumor sample for exploratory biomarker research.
9. ECOG (Eastern Oncology Cooperative Group) performance status 0-1.
10. Patient demonstrates adequate organ and marrow function within 14 days of studydrug administration:

    * Absolute neutrophil count (ANC) ≥ 1.5 × 109/L (1500/µL)
    * Lymphocyte count ≥ 0.5 × 109/L (500/µL)
    * Platelet count ≥ 75 × 109/L (75,000/µL) without transfusion
    * Hemoglobin ≥ 90 g/L (9 g/dL)
    * Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase ALP) ≤ 5 × upper limit of normal (ULN)
    * Serum bilirubin ≤ 3 × ULN
    * Serum creatinine ≤ 1.5 × ULN
    * Serum albumin ≥ 28 g/L (2.8 g/dL)
    * International normalized ratio (INR) or activated partial thromboplastin time (aPTT) ≤ 2 × ULN
11. Negative human immunodeficiency virus (HIV) test at screening
12. UA with protein less than 2+. Patients discovered to have ≥2+ proteinuria on dipstick urinalysis at baseline should undergo a 24-hour urine collection and must demonstrate <1g of protein in 24 hours.
13. Documented virology status of hepatitis, as confirmed by screening HBV and HCV tests. For patients with active HBV: HBV DNA <500 IU/mL during screening, initiation of anti-HBV treatment at least 14 days prior to first dose and willingness to continue anti-HBV treatment during the study (per local standard of care; e.g., entecavir)
14. Women of childbearing potential (WOCBP) and men with partners of child bearing potential agree to prevent pregnancy using two forms of contraception from the date of Informed Consent through 6 months after the last dose of study drug. A woman is considered to be of childbearing potential if she is postmenarchal, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries, fallopian tubes and/or uterus) or another cause as determined by the investigator (e.g., Müllerian agenesis). Per this definition, a woman with a tubal ligation is considered to be of childbearing potential. The definition of childbearing potential may be adapted for alignment with local guidelines or requirements.
15. Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not adequate methods of contraception. WOCBP potential must have a negative serum pregnancy test result within 14 days of initiating study treatment
16. WOCB must not be breastfeeding.
17. For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agreement to refrain from donating sperm, as defined below: With a female partner of childbearing potential or pregnant female partner, men must remain abstinent or use a condom during the treatment period and for 6 months after the final dose of study medication to avoid exposing the embryo. Men must refrain from donating sperm during this same period. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not adequate methods of preventing drug exposure. If required per local guidelines or regulations, information about the reliability of abstinence will be described in the local Informed Consent Form.

Exclusion Criteria:

1. Patient has been treated for this malignancy, has another active malignancy, or has had an active malignancy within the last two years.
2. Patient has fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC.
3. Patient has had a bleeding event due to untreated esophageal and/or gastric varices.
4. Patient has history of abdominal or tracheoesophageal fistula, GI perforation, or intra- abdominal abscess within 6 months of initiation of study treatment.
5. Patient has history of thrombosis, bleeding diathesis, History of Grade ≥ 4 venous thromboembolism, coagulopathy or significant vascular disease, serious, non-healing wound, active ulcer, or untreated bone fracture
6. Current or recent (< 10 days prior to initiation of study treatment) use of aspirin (> 325 mg/day), or clopidogrel (> 75 mg/day) Note: The use of full-dose oral or parenteral anticoagulants for therapeutic purpose is permitted as long as the INR and/or aPTT is within therapeutic limits (according to institution standards) within 7 days prior to initiation of study treatment and the patient has been on a stable dose of anticoagulants for ≥ 2 weeks prior to initiation of study treatment. Prophylactic use of anticoagulants is allowed. However, the use of direct oral anticoagulant therapies such as dabigatran (Pradaxa) and rivaroxaban (Xarelto) is not recommended due to bleeding risk
7. Patient has history of hemoptysis within 30 days of initiation of study treatment.
8. Patient has serious cardiac disease, such as New York Heart association Grade II or greater congestive heart failure, MI, unstable angina, etc.
9. Patient has inadequately controlled hypertension (systolic ≥ 150 mmHg and/or diastolic ≥ 100 mmHg).
10. Patient has significant pulmonary disease (tuberculosis, pneumonia, pneumonitis, etc.).
11. Patient requires recurrent drainage procedures (pleural effusion, ascites, etc.).
12. Patient has had surgical procedure within 6 weeks of initiation of study treatment.
13. Patient has history of central nervous system disease.
14. Patient has history of severe allergic/anaphylactic reactions to chimeric or humanized antibodies or fusion proteins.
15. Patient has a knownhypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab formulation.
16. Patient has known hypersensitivity to bevacizumab.
17. Patient has had any investigational agents within 28 days prior to initiation of study treatment.
18. Patient has history of severe infection within 4 weeks of initiation of treatment.
19. Patient has history of autoimmune disease or immune deficiency.
20. Patient has received a stem cell, liver, or other solid organ transplant.
21. Patient has history of other significant comorbidities that would be contraindicated for investigational treatment.
22. Patient has used:

    * High dose steroids
    * Vaccine of any kind within 4 weeks of initiating study treatment
    * Oral or IV antibiotics within 2 weeks of initiating study treatment
    * Immunostimulatory agents within 4 weeks of initiating study treatment
    * Anticoagulation therapy (aspirin permitted)
    * Total parenteral nutrition
23. Patient is pregnant or breastfeeding, or intention of becoming pregnant during study treatment or within5 months after the last dose of atezolizumab or 6 months after the last dose of atezolizumab
24. History of leptomeningeal disease
25. Uncontrolled tumor-related pain. Patients requiring pain medication must be on a stable regimen at study entry. • Symptomatic lesions (e.g., bone metastases or metastases causing nerve impingement) amenable to palliative radiotherapy should be treated prior to enrollment. Patients should be recovered from the effects of radiation. There is no required minimum recovery period. • Asymptomatic metastatic lesions that would likely cause functional deficits or intractable pain with further growth (e.g., epidural metastasis that is not currently associated with spinal cord compression) should be considered for loco-regional therapy if appropriate prior to enrollment
26. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently). Patients with indwelling catheters (e.g., PleurX) are allowed.
27. Uncontrolled or symptomatic hypercalcemia (ionized calcium ≥ 1.5 mmol/L, calcium ≥12 mg/dL or corrected serum calcium ≥ULN)
28. Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during atezolizumab treatment or within 5 months after the final dose of atezolizumab
29. Treatment with investigational therapy within 28 days prior to initiation of study treatment
30. Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies
31. Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin 2 [IL- 2]) within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to initiation of study treatment
32. Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF-α agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment, with the following exceptions:

    * Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study.
    * Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response (pCR) rate | Up to 2 years post-treatment
  Will estimate pCR rate along with the 95% credible interval.
Incidence of adverse events (AEs) | Up to 30 days post-treatment
  The AE severity grading scale for the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 will be used for assessing AE severity.

SECONDARY OUTCOMES:
Objective response rate (ORR) | At the time of surgery
  Objective response is defined as complete response or partial response, per Response Evaluation Criteria in Solid Tumors (RECIST 1.1), modified (m)RECIST1.0. ORR will be summarized along with 95% confidence intervals. Fisher's exact test will be used to correlate pCR and OR.
Duration of response (DOR) | From the date of response to the date of recurrence/disease progression, assessed up to 2 years post-treatment
  DOR will be estimated with the Kaplan-Meier methods.
Recurrence-free survival (RFS) | From the date of surgery to the date of disease recurrence or death whichever occur first, assessed up to 2 years post-treatment
  RFS will be estimated with the Kaplan-Meier methods. The log-rank test will be used to evaluate the association between pCR and RFS.
Overall survival (OS) | From the date of treatment start to the date of death or to the date of last follow-up for patients alive, assessed up to 2 years post-treatment
  OS will be estimated with the Kaplan-Meier methods. The log-rank test will be used to evaluate the association between pCR and OS.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed O Kaseb, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Houston Methodist Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: MDAndersonCancerCenter — http://www.mdanderson.org